CLINICAL TRIAL: NCT01527565
Title: A Single-Centre, Randomised, Balanced, Double-Blind, Cross-Over Trial Investigating the Bioequivalence of Two Formulations of Biphasic Insulin Aspart 70 in Healthy Male Subjects
Brief Title: Bioequivalence of Two Formulations of Biphasic Insulin Aspart 70 in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: BIASP-1489
Record Dates: First submitted 2012-02-02; First posted 2012-02-07 (Estimated); Last update posted 2017-02-24 (Actual); Status verified 2017-02

CONDITIONS: Diabetes; Healthy
MeSH Terms: conditions — Diabetes Mellitus | interventions — insulin aspart, insulin aspart protamine drug combination 30:70

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Formulation A (Experimental)
  Interventions: Drug: biphasic insulin aspart 70
- Formulation B (Experimental)
  Interventions: Drug: biphasic insulin aspart 70

INTERVENTIONS:
Drug: biphasic insulin aspart 70 — A single dose of each formulation administered subcutaneously (s.c., under the skin) on 2 dosing visits separated by a wash-out period of 6-12 days

SUMMARY:
This trial is conducted in Africa. The aim of this trial is to investigate the bioequivalence of two formulations of biphasic insulin aspart 70 in healthy male subjects.

ELIGIBILITY:
Inclusion Criteria:

* Considered generally healthy upon completion of medical history and physical
* examination, as judged by the investigator
* Body Mass Index (BMI) between 19-29 kg/m^2 (both inclusive)
* Minimum body weight of 65 kg
* Fasting blood glucose between 3.8-6.0 mmol/L
* Glycohemoglobin (HbA1c) below 6.4 %
* Non-smokers

Exclusion Criteria:

* Clinically significant abnormal hematology, biochemistry, urinalysis or ECG (electrocardiogram) screening tests, as judged by the investigator
* A history of any illness that, in the opinion of the Investigator and/or Sponsor, might confound the results of the study or pose additional risk in administering the investigational product to the subject
* History of or current addiction to alcohol or drugs of abuse as determined by the investigator (positive drug/alcohol abuse screen)
* Hepatitis B or C
* Subjects with a first-degree relative with diabetes mellitus
* Known or suspected allergy to trial product or related products
* Smoking during the past three months

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2003-01-20 (Actual); Primary Completion 2003-02-26 (Actual); Study Completion 2003-02-26 (Actual)

PRIMARY OUTCOMES:
Area under the insulin aspart curve in the interval from 0-16 hours
Cmax, maximum insulin aspart concentration

SECONDARY OUTCOMES:
tmax, the time to maximum insulin aspart concentration
Area under the insulin aspart curve
Mean residence time (MRT)
The area under the glucose infusion rate curve
GIRmax, maximum glucose infusion rate value
tGIRmax, time to maximum glucose infusion rate value
Adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Bloemfontein, South Africa

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com